CLINICAL TRIAL: NCT04638699
Title: Optimized Psycho-oncological Care Through an Interdisciplinary Care Algorithm: From Screening to Intervention
Brief Title: Optimized Psycho-oncological Care Through an Interdisciplinary Care Algorithm
Acronym: OptiScreen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Universitätsklinikum Leipzig (Other); UniversitätsKrebsCentrum Dresden (Unknown)
Responsible Party: Principal Investigator, Zimmermann, Tanja Prof. Dr., Prof. Dr. Tanja Zimmermann, Hannover Medical School
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 70113550
Record Dates: First submitted 2020-11-02; First posted 2020-11-20 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Psycho-Oncology; Visceral Cancer; Screening; Psychosocial Stressor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Survey of the actual state (No Intervention)
- Phase 2 Survey after the OptiScreen training (Other)
  Interventions: Other: OptiScreen training

INTERVENTIONS:
Other: OptiScreen training — Special psycho-oncological training for nursing staff to acquire basic knowledge about the experience of mental stress as well as diagnostics of psychosocial stress
  Arms: Phase 2 Survey after the OptiScreen training

SUMMARY:
Adequate, needs-oriented psycho-oncological care contributes to reducing the burden on cancer patients and their relatives and to improving the quality of life. There is still a need for clarification regarding the need and the determination of psychosocial needs. This multi-center study (3 centers: Hanover, Leipzig and Dresden) aims at a professionalization of psychosocial screening, in order to enable thus an exact and need-based allocation to psycho-oncological support. The optimization and professionalization of the psychosocial screening process shall be achieved by a training of oncological nursing and development of an interdisciplinary care algorithm. The aim is to examine whether "OptiScreen" increases the targeted and needs-based allocation to psycho-oncology.

DETAILED DESCRIPTION:
Adequate, needs-oriented psycho-oncological care contributes to reducing the burden on cancer patients and their families and to improving the quality of life of all those affected. In order to ensure patient-oriented psycho-oncological care, it is necessary to allocate psychologically burdened patients and patients in need of care to psycho-oncology by means of screening.

Within the framework of this multicenter study (Hannover, Leipzig and Dresden), a newly designed training of nursing staff ("OptiScreen training") on mental stress and psycho-oncological care is intended to increase the precise identification of mentally stressed patients in need of treatment, to increase the allocation of these patients to psycho-oncology and to improve interdisciplinary cooperation.

Aims of the study:

1. targeted, needs-based allocation to psycho-oncology
2. increasing the acceptance of psycho-oncological screening by patients* and treatment team
3. increase of patient competence and satisfaction
4. increasing the acceptance of psycho-oncological treatment by patients and treatment team In summary, the findings of this multi-center study should contribute to the improvement of interdisciplinary cooperation, improve the demand-oriented and targeted allocation of psychologically burdened patients to psycho-oncological care and thus develop a "best practice model" of an interdisciplinary care algorithm.

Methodology

The study will include inpatients from the visceral oncology centers at the three sites who have the necessary cognitive, physical and linguistic abilities. The study is divided into 2 phases:

Phase 1: Survey of the current status For this purpose, N = 300 patients* in the visceral oncology centers are interviewed with a questionnaire during the inpatient stay (t0) and three months later (t1).

The data collected will include psychological stress, disease management/treatment, quality of life and treatment satisfaction of persons with oncological diseases. In addition, the needs for information and support, the practicability as well as the allocation to psycho-oncological care and its utilization will be surveyed.

Execution of the "OptiScreen training": special psycho-oncological training of the nursing staff for basic knowledge about the experience of psychological stress as well as diagnostics of psychosocial stress will take place after the completion of phase 1.

Phase 2: survey after the OptiScreen training Analogous to phase 1, N = 600 patients* in the visceral oncology centers are interviewed during the inpatient stay (t0) and three months later (t1).

ELIGIBILITY:
Inclusion Criteria:

* In-patients of the visceral oncology centers at the three locations

Exclusion Criteria:

* severe physical, cognitive and/or language limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Psychological distress in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Distress Thermometer (NCCN Distress Thermometer)

SECONDARY OUTCOMES:
Frequency and extent of depression in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Patient Health Questionnaire (PHQ-9)
Frequency and extent of anxiety in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Generalized Anxiety Disorder 7 (GAD-7)
Frequency and extent of supportive care needs in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Supportive Care Needs Survey Short Form German (SCNS-SF34-G)
Frequency and extent of fear of cancer recurrence in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Progredienangstfragebogen (PA-F; Fear of Progression Questionnaire)
Frequency and changes in quality of life in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Short Form-8 Health Survey SF-8
Frequency and extent of relationship satisfaction in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Quality of Marriage Index (QMI)
Satisfaction with medical and psychosocial treatment in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  REPERES-G: Assessment of care
Frequency and extent of health competence (Access to information, understanding, evaluating and applying of information) in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  European Health Literacy Questionnaire
Frequency and extent of self-management and active patient participation in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Patient Activation Measure (PAM 13D; German version of the Patient Measure
Frequency and extent of satisfaction with body image in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Body-Image-Scale
Frequency and extent of social support in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Scales for social support during illness (SSUK Skalen zur sozialen Unterstützung bei Krankheit) zur sozialen Unterstützung bei Krankheit-8 (SSUK-8; llness-specific Social Support Scale)
Frequency and extent of resources (Health promoting activities, active participation, emotional stress, self-monitoring etc.in cancer patients (CG vs. IG) and changes over time | T0 (at hospital stay) and T1 (3 months later)
  Health Education Impact Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Zimmermann, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided